CLINICAL TRIAL: NCT02397629
Title: Using Serum Parathyroid Hormones and Calcium to Improve Prostate Cancer Diagnosis
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00014769; CCCWFU 85B10 (Other: Wake Forest University Health Sciences)
Record Dates: First submitted 2015-03-17; First posted 2015-03-25 (Estimated); Last update posted 2022-03-11 (Actual); Status verified 2018-07

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples for measurement of PTHrP
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients Undergoing Prostate Biopsy: Men referred for biopsy because of an abnormal or suspicious PSA digital rectal exam, or both.
  Interventions: Other: This study has no intervention

INTERVENTIONS:
Other: This study has no intervention

SUMMARY:
This is a cross sectional study to examine the relationship between serum calcium and PTHrP and serum PSA in men referred for prostate biopsy at Wake Forest University.

DETAILED DESCRIPTION:
This is a cross sectional study to examine the relationship between serum calcium and PTHrP and serum PSA in men referred for prostate biopsy at Wake Forest University. Men scheduled for biopsy will be approached by the study nurse who will explain the study and invite the men to participate. After the patients provide written consent, she/he will obtain the following information from the patient chart: age, race (self-report, white, black, other), height, weight (for determination of Body Mass Index, a variable reported to influence PSA). Blood draw for study analytes will be coordinated with routine blood draw for PSA testing to minimize the need for an additional needle stick. A copy of the informed consent is given to the patient and the original is placed in a file for the P.I.

The biopsy status of men at the time they are invited to participate is unknown. Men are "sorted" into cancer and non-cancer groups only after their biopsies are read. Serum samples are sent to the Department of Laboratory Medicine at Wake Forest. All assays are performed "in house". Based on consultation with our urologists, we anticipate that approximately 30% of the biopsies will be positive (i.e., prostate cancer). The majority (approximately 70%) will be negative (benign). Approximately 1-2% of the biopsies may be classified as "indeterminate". Because there will not be a sufficient number of "indeterminate" pathologies to be treated as a separate category, this group will not be analyzed further. However, men with "indeterminate" biopsies are eligible for the study if they are re-biopsied.

ELIGIBILITY:
Inclusion Criteria:

* Men age > 40 years
* Men referred for biopsy because of an abnormal or suspicious PSA digital rectal exam, or both.
* Ability and willingness to sign a written, IRB-approved informed consent document

Exclusion Criteria:

* Men using drugs known to interfere with serum PSA or with serum PTHrP and calcium. Drugs known to interfere with PSA include 5-alpha-reductase inhibitors (Proscar). Drugs known to interfere with calcium and/or PTH include lithium and thiazide diuretics.
* Patients with prior transurethral resection of the prostate (TURP) or equivalent procedure (laser incision). In these men the reduction in prostatic volume may give a biased estimate of the relationship between PSA, calcium and PTHrP.
* Patients on dialysis. These are excluded because dialysis increases the percentage of free PSA in serum.

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men > 40 years old scheduled for a prostate biopsy
Sampling Method: Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2013-05; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
To measure the relationship of calcium and PTH levels to PSA levels in patients receiving a prostate biopsy. | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Ram Pathak, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Comprehensive Cancer Center of Wake Forset University, Winston-Salem, North Carolina, United States